CLINICAL TRIAL: NCT05120817
Title: Me or We? Emphasizing the Personal Versus the Social in Educational Interventions For Decreasing Vaccine Hesitancy
Brief Title: Emphasizing the Personal Versus the Social in Educational Interventions For Decreasing Vaccine Hesitancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Research University Higher School of Economics (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hsestudy2021
Record Dates: First submitted 2021-11-02; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Vaccine Hesitancy; Communication
Keywords: vaccine hesitancy; education; COVID-19 vaccine
MeSH Terms: conditions — Vaccination Hesitancy; Communication | interventions — Social Work

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention): Participants do not undergo any intervention. Pre-and post data collection only.
- Personal (Experimental): Participants are exposed to the message about the personal benefits (and costs) of vaccination which refers to their own safety, their freedoms, their worries about the well-being of their significant others.
  Interventions: Behavioral: "Personal" intervention
- Social (Experimental): Participants are exposed to the message about the social benefits (and costs) of vaccination which refers to public safety, the well-being of others in their community, the vulnerable groups, etc.
  Interventions: Behavioral: "Social" intervention
- Personal + Social (Experimental): Participants are exposed to the message about both personal and social benefits (and costs) of vaccination. The message alludes to personal safety as well as public safety and the strain on the healthcare system associated with the uncontrollable spread of the virus.
  Interventions: Behavioral: "Personal" + "Social" intervention

INTERVENTIONS:
Behavioral: "Personal" intervention — Participants will receive a link with an invitation to watch a 10-minute educational video about the personal benefits and costs of vaccination against COVID-19. They will also go through pre-and post-test data collection.
  Arms: Personal
Behavioral: "Social" intervention — Participants will receive a link with an invitation to watch a 10-minute educational video about the social benefits and costs of vaccination against COVID-19. They will also go through pre-and post-test data collection.
  Arms: Social
Behavioral: "Personal" + "Social" intervention — Participants will receive a link with an invitation to watch a 10-minute educational video about both personal and social benefits and costs of vaccination against COVID-19. They will also go through pre-and post-test data collection.
  Arms: Personal + Social

SUMMARY:
This experimental study aims to investigate the effect of different types of educational interventions on overcoming Coronavirus disease 2019 (COVID-19) vaccine hesitancy among the Higher School of Economics (HSE) bachelor students in Russia.

DETAILED DESCRIPTION:
The researchers aim to investigate the effectiveness of three types of educational interventions on overcoming COVID-19 vaccine hesitancy among the HSE bachelor students. The study design implies the comparison of three types of educational interventions which differ in the message that they deliver to the participants: the personal, the social, and a combination of the two. The effects of these interventions will be compared to the control group with no intervention.

Participants in these three experimental groups will receive a link to an educational video about the benefits and costs of vaccination against COVID-19. The videos for the three groups will contain information about vaccination, but each of them will have a different focus.

The participants will be hired on a voluntary basis. All the participants will sign the informed consent form, and the measures will be taken to ensure that their personal data will be protected.

ELIGIBILITY:
Inclusion Criteria:

* HSE bachelor students from 18 to 25 years old, who agreed to participate in the study.

Exclusion Criteria:

* Students who have got vaccinated already.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4000 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Real vaccination status | 1-3 months
  Participants report whether they have got vaccinated against COVID-19.

SECONDARY OUTCOMES:
Knowledge, attitudes, and self-reported behaviors | 1-3 months
  Participants will be given a questionnaire to test their knowledge, attitudes towards vaccination, and self-reported behaviors surrounding vaccination and safety protocols. The questionnaire will be designed by the researchers.

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Loyalka, PhD, Study Chair — Stanford University
Locations (1):
- Higher School of Economics, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
The deidentified individual participant data (IPD) collected in the course of the experiment will be made available. The Study Protocol, Statistical Analysis Plan, and Informed Consent Form will also be available.
  All data will be available on request after 6 months following article publication.
Supporting Information: Study Protocol, Analytic Code
Time Frame: 6 months following article publication
Access Criteria: The IPD will be shared upon request with a sound description of the intended study.